CLINICAL TRIAL: NCT00353223
Title: Interpersonal Psychotherapy for Depression in Patients With Heart Failure
Brief Title: Interpersonal Psychotherapy for Depression in People With Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R34MH073566 (NIH); R34MH073566 (NIH); DATR A4-GPS
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Depression; Heart Failure, Congestive
Keywords: Heart Failure; Functional Impairment; Health-Related Quality of Life; Telemedicine
MeSH Terms: conditions — Depression; Heart Failure | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Participants will receive combined interpersonal and behavioral psychotherapy aimed at reducing depression in patients with heart failure.
  Interventions: Behavioral: Interpersonal and behavioral psychotherapy
- B (Active Comparator): Participants will receive the attention control condition.
  Interventions: Behavioral: Attention control (AC) condition

INTERVENTIONS:
Behavioral: Interpersonal and behavioral psychotherapy — Participants will receive a combined intervention of interpersonal and behavioral psychotherapy designed for people with heart failure. Participants will attend 12 sessions, 9 of which will be 30-minute to 1-hour sessions over the phone. The remaining 3 will be in-home visits, lasting 1 to 2 hours. The psychotherapy sessions will allow participants to discuss how they are coping with their illness and loss of functioning. They will also aim to help participants with heart failure to develop new recreational activities in keeping with their new level of functioning.
  Arms: A
Behavioral: Attention control (AC) condition — The AC group will not receive therapy. Instead, a clinician will ask them questions about their depression and heart failure. Participants will attend 12 sessions, 9 of which will be 30-minute to 1-hour sessions over the phone. The remaining 3 will be in-home visits, lasting 1 to 2 hours.
  Arms: B

SUMMARY:
This study will evaluate the effectiveness of interpersonal psychotherapy and behavioral activation techniques in treating depression in people with congestive heart failure.

DETAILED DESCRIPTION:
This study aims to develop an intervention based on interpersonal psychotherapy (IPT) and behavioral activation (BA) techniques to treat depression in people with congestive heart failure. By addressing how participants' loss of functioning has changed their personal relationships, the psychotherapy will help participants to discuss how they are coping with their illness and loss of functioning. It will also help participants with heart failure to develop new recreational activities in keeping with their new level of functioning. The study will first develop the methods for the intervention and then pilot the study in a small randomized, controlled trial.

Access to care has been a major barrier to treatment in prior psychosocial studies in cardiac patients. Because many people with advanced heart failure are homebound, the treatment in this study will be administered primarily by telephone, which will greatly enhance dissemination of the intervention. The treatment techniques developed will be applicable to a range of homebound patients and frail elderly, not just patients with heart failure. The long-term goal of the study is to develop pragmatic interventions to reduce depression in people coping with irreversible functional decline.

Specific Aim #1 - Treatment Standardization: The purpose of this phase will be to develop an intervention that addresses the emotional and behavioral consequences of heart failure by 1) integrating IPT and BA techniques to address both interpersonal and functional issues related to disability, 2) applying IPT theory of "role transition" and "grief and loss" to coping with functional decline, 3) applying BA interventions to maximize functioning in patients with severe impairment due to medical illness, 4) developing the techniques needed to implement both IPT and BA successfully over the telephone, 5) developing the methods to implement an appropriate attention control (AC) group, 6) generating complementary visual materials for patients to enhance understanding of the therapeutic model, and 7) evaluating a range of functional assessments to be used as alternative outcomes. Two therapists will conduct the treatment by telephone with 15 depressed heart failure patients. Participants' baseline 17-item Hamilton Rating Scale for Depression (HRSD) total score will be compared with the HRSD total score from Weeks 6 and 12.

Specific Aim #2 - Treatment Evaluation: The purpose of this phase will be to pilot the new treatment in a randomized, controlled trial of people suffering major or minor depression. This phase will include the application of therapist training techniques, assessment of treatment fidelity, and selection of optimal outcome, adherence, process, and treatment quality measures. Participants will be randomly assigned to receive IPT or an attention control condition (AC). Both groups will attend 12 sessions, 9 of which will be 30-minute to 1-hour sessions over the phone. The remaining 3 will be in-home visits lasting 1 to 2 hours. The IPT group will receive IPT designed for people with heart failure. The AC group will not receive therapy. Instead, a clinician will ask them questions about their depression and heart failure. Depressive symptoms will be measured for all participants using the HRSD at baseline and Weeks 6 and 12.

Specific Aim #3 - Treatment Feasibility: In both the standardization and evaluation phases, specific treatment feasibility issues will be addressed. The main feasibility issue will be the acceptability and effectiveness of a telephone administered intervention with severely impaired older people. In addition, recruitment and retention issues will be addressed in all stages of treatment development. The main outcome of this aim will be adequate recruitment sources, including adequate representation of minorities, to conduct a large scale R01 intervention.

ELIGIBILITY:
Inclusion Criteria:

* Current heart failure
* Current minor or major depression
* Score of 14 or higher on the Beck Depression Inventory-II

Exclusion Criteria:

* Score of less than 24 on the Mini-Mental State Exam

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Score on the 17-item HRSD | Measured at Week 12

SECONDARY OUTCOMES:
Health-related quality of life | Measured at Week 12
Interpersonal functioning | Measured at Week 12
Behavioral activation | Measured at Week 12
Self care of heart failure | Measured at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L. Turvey, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States